CLINICAL TRIAL: NCT06225947
Title: A Prospective, Multi-center, 3-month, Observational Study to Evaluate the Effectiveness and Safety of Lemborexant in Chinese Patients With Insomnia in Real World Setting.
Brief Title: Patient-Reported Outcomes for Lemborexant in Chinese Participants With Insomnia
Acronym: PROEM
Status: Recruiting | Type: Observational
Sponsor: Guangdong Provincial People's Hospital (Other)
Collaborators: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: KY2023-1072-02
Record Dates: First submitted 2024-01-17; First posted 2024-01-26 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-02

CONDITIONS: Insomnia
Keywords: insomnia; lemborexant
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — lemborexant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Lemborexant(LEM): Subjects will be administered with Lemborexant(LEM). The dosage of LEM is 5 mg or 10mg taken no more than once per night during the study.
  Interventions: Drug: Lemborexant 5 MG

INTERVENTIONS:
Drug: Lemborexant 5 MG — The recommended dosage of Lemborexant(LEM) is 5 mg taken no more than once per night, immediately before going to bed, with at least 7 hours remaining before the planned time of awakening. The dose may be increased to the maximum recommended dose of 10 mg based on clinical response and tolerability.
  Other Names: DAYVIGO

SUMMARY:
This study is a prospective, open-label, single arm, multicenter study lasting 12 weeks to evaluate effectiveness and safety of lemborexant(LEM). Patient self-evaluation reports and safety events will be collected at baseline and 4 visits during treatment.

DETAILED DESCRIPTION:
This study is a prospective, open-label, single arm, multicenter study lasting 12 weeks to evaluate effectiveness and safety of lemborexant(LEM). Adult patients diagnosed with insomnia (including chronic and short-term insomnia) in the fifth edition of the Diagnostic and Statistical Manual of Mental Disorders (DSM-5) and ISI ≥10, clinically judged to need pharmacological treatment will be enrolled.Patients will be administered with LEM, and patient self-evaluation reports and safety events will be collected at baseline and each visit during treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years) and agreed to participate in the study, regardless of gender.
* Diagnosed with insomnia according to DSM-5.
* Insomnia Severity Index (ISI) score >10.
* Subjects who can guarantee at least 7 hours of bedtime.
* Subjects signed informed consent forms after the prescription.

Exclusion Criteria:

* Beings unable to understand the questionnaire.
* PHQ-9 scores ≥ 20.
* GAD-7 scores ≥ 15.
* Suicidal thoughts/behaviors in the past one month or history of suicide, etc.
* Severe psychiatric disorder in the judgment of the investigator prevents completion of the trial.
* History of serious illness, mental illness, medication use, and uncontrolled poor sleep habits that the investigator believes interfere with the study evaluation or the safety of the subject.
* According to the precautions listed in the instructions, there are any contraindications or other conditions for which the use is prohibited (such as narcolepsy, severe liver damage, pregnant, nursing or pregnant women, etc.).
* Other conditions not considered appropriate for participation by clinicians.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese patients with insomnia administered with LEM.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-02-22 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with insomnia remission | Baseline, week 1, week 2, week 4, week 12
  Percentage of patients with total ISI score below 8 points after Lemborexant treatment. Insomnia remission is defined as total ISI below 8points. The ISI is a 7-item self-report questionnaire assessing the nature, severity and impact of insomnia. A 5-point likert scale is used to rate each item, score range=0 ~28. Higher score indicate worse severity.

SECONDARY OUTCOMES:
Retention rate of Lemborexant treatment at each visit | up to week 12
  The retention rate is defined as the percentage of participants remaining on Lemborexant treatment regardless of treatment pattern, starting from the first dose of study drug.
  The retention is primarily defined as follows:
  * Patients who wish to continue LEM treatment at each visit.
  * Patients who wish to continue LEM treatment at each visit. but do not actually continue with a reason not related to the efficacy or safety of LEM treatment (including, but not limited to relocation, clinic transfer, or a burden of site visit expenses)
Change from baseline of mean ISI score at each visit | Baseline, week 1, week 2, week 4, week 12
  Change of mean ISI score from baseline was defined as the average score of ISI scale at each visit relative to baseline. The ISI is a 7-item self-report questionnaire assessing the nature, severity and impact of insomnia. A 5-point likert scale is used to rate each item, score range=0 ~28. Higher score indicate worse severity.
Change from baseline of mean ISI score at LEM 5mg and 10 mg at each visit | Baseline, week 1, week 2, week 4, week 12
  Change of mean ISI score from baseline was defined as the average score of ISI scale at LEM 5mg and LEM 10mg at each visit relative to baseline. The ISI is a 7-item self-report questionnaire assessing the nature, severity and impact of insomnia. A 5-point likert scale is used to rate each item, score range=0 ~28. Higher score indicate worse severity.
Change from baseline of mean ISI score at age <55 and ≥ 55 at each visit | Baseline, week 1, week 2, week 4, week 12
  Change of mean ISI score from baseline was defined as the average score of ISI scale at age <55 and ≥ 55 at each visit relative to baseline. The ISI is a 7-item self-report questionnaire assessing the nature, severity and impact of insomnia. A 5-point likert scale is used to rate each item, score range=0 ~28. Higher score indicate worse severity.
Change from baseline of mean ISI score with LEM monotherapy, alternative therapy, and combination therapy at each visit | Baseline, week 1, week 2, week 4, week 12
  Change of mean ISI score from baseline was defined as the average score of ISI scale with LEM monotherapy, alternative therapy, and combination therapy at each visit relative to baseline.
  * LEM monotherapy is defined as participant who has not previously taken hypnotics(e.g. benzodiazepine receptor agonists, sedative antidepressants, etc.) and initiated of LEM monotherapy.
  * Alternative therapy is defined as participant who discontinued benzodiazepine hypnotics with initiation of LEM.
  * Combination therapy is defined as participant who add LEM to the current medication of benzodiazepine hypnotics.
  The ISI is a 7-item self-report questionnaire assessing the nature, severity and impact of insomnia. A 5-point likert scale is used to rate each item, score range=0 ~28. Higher score indicate worse severity.
Change from baseline of mean ISI score in patients with depression symptoms at each visit | Baseline, week 1, week 2, week 4, week 12
  Change of mean ISI score from baseline was defined as the average score of ISI scale in patients with depression symptoms at each visit relative to baseline.
  The ISI is a 7-item self-report questionnaire assessing the nature, severity and impact of insomnia. A 5-point likert scale is used to rate each item, score range=0 ~28. Higher score indicate worse severity.
  Patients with depression symptoms were defined as patients with PHQ-9 ≥ 10. The PHQ-9 is a 9-items self-report questionnaire assessing depression and severity. A 4-point likert scale is used to rate each item, score range=0-27, with higher scores indicating greater severity of depression.
Proportion of insomnia treatment responders at each visit | Baseline, week 4, week 12
  Responder was defined as total ISI reduction≥6 compared to baseline. The ISI is a 7-item self-report questionnaire assessing the nature, severity and impact of insomnia. A 5-point likert scale is used to rate each item, score range=0 ~28. Higher score indicate worse severity.
Changes of mean ESS score at each visit | Baseline, week 1, week 2, week 4, week 12
  Change of mean ESS score from baseline was defined as the average score of ESS scale at each visit relative to baseline.The ESS is a 8-items self-report questionnaire assessing daytime sleepiness. A 4-point likert scale is used to rate each item, score range=0-24, with higher scores indicating greater daytime sleepiness.
Changes of mean ESS score at LEM 5mg and 10mg at each visit | Baseline, week 1, week 2, week 4, week 12
  Change of mean ESS score from baseline was defined as the average score of ESS scale at LEM 5mg and 10 mg at each visit relative to baseline.The ESS is a 8-items self-report questionnaire assessing daytime sleepiness. A 4-point likert scale is used to rate each item, score range=0-24, with higher scores indicating greater daytime sleepiness.
Changes of mean ESS score at age <55 and ≥ 55 at each visit | Baseline, week 1, week 2, week 4, week 12
  Change of mean ESS score from baseline was defined as the average score of ESS scale at age <55 and ≥ 55 at each visit relative to baseline.The ESS is a 8-items self-report questionnaire assessing daytime sleepiness. A 4-point likert scale is used to rate each item, score range=0-24, with higher scores indicating greater daytime sleepiness.
Changes of mean ESS score with LEM monotherapy, alternative therapy, and combination therapy at each visit | Baseline, week 1, week 2, week 4, week 12
  Change of mean ESS score from baseline was defined as the average score of ESS scale with LEM monotherapy, alternative therapy, and combination therapy at each visit relative to baseline.
  * LEM monotherapy is defined as participant who has not previously taken hypnotics(e.g. benzodiazepine receptor agonists, sedative antidepressants, etc.) and initiated of LEM monotherapy.
  * Alternative therapy is defined as participant who discontinued benzodiazepine hypnotics with initiation of LEM.
  * Combination therapy is defined as participant who add LEM to the current medication of benzodiazepine hypnotics.
  The ESS is a 8-items self-report questionnaire assessing daytime sleepiness. A 4-point likert scale is used to rate each item, score range=0-24, with higher scores indicating greater daytime sleepiness.
Changes of mean ESS score in patients with depression symptoms at each visit | Baseline, week 1, week 2, week 4, week 12
  Change of mean ESS score from baseline was defined as the average score of ESS scale in patients with depression symptoms at each visit relative to baseline.
  The ESS is a 8-items self-report questionnaire assessing daytime sleepiness. A 4-point likert scale is used to rate each item, score range=0-24, with higher scores indicating greater daytime sleepiness.
  Patients with depression symptoms were defined as patients with PHQ-9 ≥ 10. The PHQ-9 is a 9-items self-report questionnaire assessing depression and severity. A 4-point likert scale is used to rate each item, score range=0-27, with higher scores indicating greater severity of depression.
Changes of mean QOL-BREF score at each visit | Baseline, week 4, week 12
  Change of mean QOL-BREF score from baseline was defined as the average score of QOL-BREF scale at each visit relative to baseline. QOL-BREF is used 26-items WHOQOL-BREF assessing quality of life. A 5-point likert scale is used to rate each item, score range=0-100. It yields a multi-dimensional profile of scores across domains and sub-domains (facets) of quality of life.
Changes of mean QOL-BREF score at LEM 5mg and 10mg at each visit | Baseline, week 4, week 12
  Change of mean QOL-BREF score from baseline was defined as the average score of QOL-BREF scale at LEM 5mg and 10mg at each visit relative to baseline. QOL-BREF is used 26-items WHOQOL-BREF assessing quality of life. A 5-point likert scale is used to rate each item, score range=0-100. It yields a multi-dimensional profile of scores across domains and sub-domains (facets) of quality of life.
Changes of mean QOL-BREF score at age <55 and ≥ 55 at each visit | Baseline, week 4, week 12
  Change of mean QOL-BREF score from baseline was defined as the average score of QOL-BREF scale at age <55 and ≥ 55 at each visit relative to baseline. QOL-BREF is used 26-items WHOQOL-BREF assessing quality of life. A 5-point likert scale is used to rate each item, score range=0-100. It yields a multi-dimensional profile of scores across domains and sub-domains (facets) of quality of life.
Changes of mean QOL-BREF score with LEM monotherapy, alternative therapy, and combination therapy at each visit | Baseline, week 4, week 12
  Change of mean QOL-BREF score from baseline was defined as the average score of QOL-BREF scale with LEM monotherapy, alternative therapy, and combination therapy at each visit relative to baseline.
  * LEM monotherapy is defined as participant who has not previously taken hypnotics(e.g. benzodiazepine receptor agonists, sedative antidepressants, etc.) and initiated of LEM monotherapy.
  * Alternative therapy is defined as participant who discontinued benzodiazepine hypnotics with initiation of LEM.
  * Combination therapy is defined as participant who add LEM to the current medication of benzodiazepine hypnotics.
  QOL-BREF is used 26-items WHOQOL-BREF assessing quality of life. A 5-point likert scale is used to rate each item, score range=0-100. It yields a multi-dimensional profile of scores across domains and sub-domains (facets) of quality of life.
Changes of mean QOL-BREF score in patients with depression symptoms at each visit | Baseline, week 4, week 12
  Change of mean QOL-BREF score from baseline was defined as the average score of QOL-BREF scale in patients with depression symptoms at each visit relative to baseline.
  QOL-BREF is used 26-items WHOQOL-BREF assessing quality of life. A 5-point likert scale is used to rate each item, score range=0-100. It yields a multi-dimensional profile of scores across domains and sub-domains (facets) of quality of life.
  Patients with depression symptoms were defined as patients with PHQ-9 ≥ 10. The PHQ-9 is a 9-items self-report questionnaire assessing depression and severity. A 4-point likert scale is used to rate each item, score range=0-27, with higher scores indicating greater severity of depression.
Changes of mean PHQ-9 score at each visit | Baseline, week 1, week 2, week 4, week 12
  Change of mean PHQ-9 score from baseline was defined as the average score of PHQ-9 scale at each visit relative to baseline. The PHQ-9 is a 9-items self-report questionnaire assessing depression and severity. A 4-point likert scale is used to rate each item, score range=0-27, with higher scores indicating greater severity of depression.
Changes of mean PHQ-9 score at LEM 5mg and 10mg at each visit | Baseline, week 1, week 2, week 4, week 12
  Change of mean PHQ-9 score from baseline was defined as the average score of PHQ-9 scale at LEM 5mg and 10mg at each visit relative to baseline. The PHQ-9 is a 9-items self-report questionnaire assessing depression and severity. A 4-point likert scale is used to rate each item, score range=0-27, with higher scores indicating greater severity of depression.
Changes of mean PHQ-9 score at age <55 and ≥ 55 at each visit | Baseline, week 1, week 2, week 4, week 12
  Change of mean PHQ-9 score from baseline was defined as the average score of PHQ-9 scale at age <55 and ≥ 55 at each visit relative to baseline. The PHQ-9 is a 9-items self-report questionnaire assessing depression and severity. A 4-point likert scale is used to rate each item, score range=0-27, with higher scores indicating greater severity of depression.
Changes of mean PHQ-9 score with LEM monotherapy, alternative therapy, and combination therapy at each visit | Baseline, week 1, week 2, week 4, week 12
  Change of mean PHQ-9 score from baseline was defined as the average score of PHQ-9 scale with LEM monotherapy, alternative therapy, and combination therapy at each visit relative to baseline.
  * LEM monotherapy is defined as participant who has not previously taken hypnotics(e.g. benzodiazepine receptor agonists, sedative antidepressants, etc.) and initiated of LEM monotherapy.
  * Alternative therapy is defined as participant who discontinued benzodiazepine hypnotics with initiation of LEM.
  * Combination therapy is defined as participant who add LEM to the current medication of benzodiazepine hypnotics.
  The PHQ-9 is a 9-items self-report questionnaire assessing depression and severity. A 4-point likert scale is used to rate each item, score range=0-27, with higher scores indicating greater severity of depression.
Changes of mean PHQ-9 score in patients with depression symptoms at each visit | Baseline, week 1, week 2, week 4, week 12
  Change of mean PHQ-9 score from baseline was defined as the average score of PHQ-9 scale in patients with depression symptoms at each visit relative to baseline.
  Patients with depression symptoms were defined as patients with PHQ-9 ≥ 10.The PHQ-9 is a 9-items self-report questionnaire assessing depression and severity. A 4-point likert scale is used to rate each item, score range=0-27, with higher scores indicating greater severity of depression.
Changes of mean GAD-7 score at each visit | Baseline, week 1, week 2, week 4, week 12
  Change of mean GAD-7 score from baseline was defined as the average score of GAD-7 scale at each visit relative to baseline. The GAD-7 is a 7-items self-reported questionnaire assessing anxiety disorder severity. A 4-point likert scale is used to rate each item, score range=0-21, with higher scores indicating greater severity of anxiety.
Changes of mean GAD-7 score at LEM 5mg and 10mg at each visit | Baseline, week 1, week 2, week 4, week 12
  Change of mean GAD-7 score from baseline was defined as the average score of GAD-7 scale at LEM 5mg and 10mg at each visit relative to baseline. The GAD-7 is a 7-items self-reported questionnaire assessing anxiety disorder severity. A 4-point likert scale is used to rate each item, score range=0-21, with higher scores indicating greater severity of anxiety.
Changes of mean GAD-7 score at age <55 and ≥ 55 at each visit | Baseline, week 1, week 2, week 4, week 12
  Change of mean GAD-7 score from baseline was defined as the average score of GAD-7 scale at age <55 and ≥ 55 at each visit relative to baseline. The GAD-7 is a 7-items self-reported questionnaire assessing anxiety disorder severity. A 4-point likert scale is used to rate each item, score range=0-21, with higher scores indicating greater severity of anxiety.
Changes of mean GAD-7 score with LEM monotherapy, alternative therapy, and combination therapy at each visit | Baseline, week 1, week 2, week 4, week 12
  Change of mean GAD-7 score from baseline was defined as the average score of GAD-7 scale with LEM monotherapy, alternative therapy, and combination therapy at each visit relative to baseline.
  * LEM monotherapy is defined as participant who has not previously taken hypnotics(e.g. benzodiazepine receptor agonists, sedative antidepressants, etc.) and initiated of LEM monotherapy.
  * Alternative therapy is defined as participant who discontinued benzodiazepine hypnotics with initiation of LEM.
  * Combination therapy is defined as participant who add LEM to the current medication of benzodiazepine hypnotics.
  The GAD-7 is a 7-items self-reported questionnaire assessing anxiety disorder severity. A 4-point likert scale is used to rate each item, score range=0-21, with higher scores indicating greater severity of anxiety.
Changes of mean GAD-7 score in patients with depression symptoms at each visit | Baseline, week 1, week 2, week 4, week 12
  Change of mean GAD-7 score from baseline was defined as the average score of GAD-7 scale in patients with depression symptoms at each visit relative to baseline.
  The GAD-7 is a 7-items self-reported questionnaire assessing anxiety disorder severity. A 4-point likert scale is used to rate each item, score range=0-21, with higher scores indicating greater severity of anxiety.
  Patients with depression symptoms were defined as patients with PHQ-9 ≥ 10. The PHQ-9 is a 9-items self-report questionnaire assessing depression and severity. A 4-point likert scale is used to rate each item, score range=0-27, with higher scores indicating greater severity of depression.
Incidence of Treatment-Emergent Adverse Events during LEM treatment | Up to week 12
  Percentage of Participants Reporting one or More Treatment-emergent Adverse Events (TEAEs), TEAEs Leading to Discontinuation, and TEAEs by Severity
Incidence of Serious Adverse Events during LEM treatment | Up to week 12
  Percentage of Participants Reporting one or More Serious Adverse Events (SAEs)

CONTACTS AND LOCATIONS:
Overall Officials: Fujun Jia, MD, Principal Investigator — Guangdong Provincial People's Hospital; Bin Zhang, MD, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (5):
- China (5):
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Sun Yat-sen Memorial Hospital, Guangzhou, Guangdong
  - Guangzhou United Family Hospital, Guangzhou, Guangdong
  - Nanfang Hospital, Guangzhou, Guangdong
  - Clifford Hospital, Guangzhou, Guangdong

IPD SHARING:
Plan to Share IPD: No